CLINICAL TRIAL: NCT01984632
Title: Single-port Laparoscopic Myomectomy Using Barbed Suture Versus Multi-port One: a Multi-center Randomized Controlled Trial
Brief Title: Barbed Suture in Single-port Laparoscopic Myomectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYO04
Record Dates: First submitted 2013-11-03; First posted 2013-11-15 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Uterine Myoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-port laparoscopic myomectomy (Experimental): We will use barbed suture (V-Loc) under intervention of single-port laparoscopic myomectomy
  Interventions: Procedure: Single-port laparoscopic myomectomy
- Multi-port laparoscopic myomectomy (Active Comparator): We will use barbed suture(V-Loc) under intervention of multi-port laparoscopic myomectomy.
  Interventions: Procedure: Multi-port laparoscopic myomectomy

INTERVENTIONS:
Procedure: Single-port laparoscopic myomectomy — The aim of this study is to compare single-port laparoscopic myomectomy using barbed suture (experimental group) with multi-port laparoscopic myomectomy using barbed suture (control group) in terms of operative time (esp. suturing time).
  Arms: Single-port laparoscopic myomectomy
Procedure: Multi-port laparoscopic myomectomy — The aim of this study is to compare single-port laparoscopic myomectomy using barbed suture (experimental group) with multi-port laparoscopic myomectomy using barbed suture(control group) in terms of operative time (esp. suturing time).
  Arms: Multi-port laparoscopic myomectomy

SUMMARY:
The aim of this study is to test our hypothesis that the use of unidirectional knotless barbed suture in single-port laparoscopic myomectomy could facilitate the suture of uterine wall defect after myoma enucleation as multi-port laparoscopic myomectomy did.

DETAILED DESCRIPTION:
The investigators plan to perform a multi-center randomized clinical trial on women scheduled for laparoscopic myomectomy. All women will get the same preoperative and postoperative care. Women will be assigned by chance to one of two groups: one group will receive single-port laparoscopic myomectomy using V-Loc™ suture material (study group). The other group will receive conventional multi-port laparoscopic myomectomy using V-Loc™ suture material (control group). The investigators will collect information on suturing time and complications related to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Image-confirmed uterine myoma
* Number of myoma ≤2 and largest size ≤10cm
* Women who were scheduled to have laparoscopic myomectomy
* Appropriate medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification 1 or 2)

Exclusion Criteria:

* Women with pedunculated subserosal myoma or submucosal myoma
* Women undergoing concomitant complex surgical procedures at the time of laparoscopic myomectomy such as severe adhesiolysis or resection for severe endometriosis
* Women with any suggestion of malignant uterine or adnexal diseases
* Women with diabetics, malignancy, or malnutrition, which can affect wound healing
* Women having major medical comorbidity or psychiatric illness, which could affect follow-up and/or compliance
* Women who refuse to participate or give consent to the procedures

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Suturing time | Intra-operative
  the time duration for the suture of uterine wall defect after myoma enucleation during laparoscopic myomectomy

SECONDARY OUTCOMES:
Cosmetic satisfaction | Post-surgery 1 month and 3 month
  We will compare patient's cosmetic satisfaction through self-reported questionnaire (Body image Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD, Principal Investigator — CHA Gangnam Medical Center, CHA university, Seoul, Republic of Korea
Locations (4):
- South Korea (4):
  - National Health Insurance Service Ilsan Hospital, Goyang
  - CHA Gangnam Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Song T, Kim TJ, Lee SH, Kim TH, Kim WY. Laparoendoscopic single-site myomectomy compared with conventional laparoscopic myomectomy: a multicenter, randomized, controlled trial. Fertil Steril. 2015 Nov;104(5):1325-31. doi: 10.1016/j.fertnstert.2015.07.1137. Epub 2015 Aug 8. PMID 26263079